CLINICAL TRIAL: NCT05671029
Title: A Double-blind, Single-center, Randomized, Placebo- and Positive-controlled, Parallel-group Trial With a Nested Crossover Part on the Electrocardiographic Effects 100 and 400 mg Pritelivir Per Day in Healthy Subjects: a Thorough QT/QTc Trial
Brief Title: Thorough QT/QTc of Pritelivir in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AiCuris Anti-infective Cures AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AIC316-03-I-07
Record Dates: First submitted 2022-12-12; First posted 2023-01-04 (Actual); Results first posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-02

CONDITIONS: Healthy Subjects
Keywords: Pritelivir, QT, QTc, thorough QT study
MeSH Terms: interventions — pritelivir; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Subjects (32 male and female subjects) received 400 mg pritelivir on Day 1, 100 mg pritelivir from Day 2 to 6 and 400 mg pritelivir from Day 7 to 16.
  Furthermore, these subjects received moxifloxacin matching placebo on the Days 2 and 17.
  Interventions: Drug: Pritelivir and moxifloxacin placebo
- Group 2a (Experimental): Subjects (16 male and female subjects) received the respective amounts of tablets of matching pritelivir matching placebo on Day 1 to Day 16 in Group 2a as verum tablets in Group1.
  Furthermore, these subjects received 400 mg moxifloxacin on Day 2 and moxifloxacin matching placebo on Day 17.
  Interventions: Drug: Pritelivir placebo, moxifloxacin and moxifloxacin placebo
- Group 2b (Experimental): Subjects (16 male and female subjects) received the respective amounts of tablets of matching pritelivir matching placebo on Day 1 to Day 16 in Group 2b as verum tablets in Group1.
  Furthermore, these subjects received moxifloxacin matching placebo on Day 2 and 400 mg moxifloxacin on Day 17.
  Interventions: Drug: Pritelivir placebo, moxifloxacin placebo and moxifloxacin

INTERVENTIONS:
Drug: Pritelivir and moxifloxacin placebo — oral administration
  Arms: Group 1
Drug: Pritelivir placebo, moxifloxacin and moxifloxacin placebo — oral administration
  Arms: Group 2a
Drug: Pritelivir placebo, moxifloxacin placebo and moxifloxacin — oral administration
  Arms: Group 2b

SUMMARY:
This Phase 1 clinical trial was a double-blind, single-center, randomized and placebo-controlled trial in which healthy male and female subjects received in 2 parallel-groups daily oral doses of pritelivir (Group 1) or matching placebo (Group 2). Within Group 2, a single oral administration of moxifloxacin (positive control) and corresponding matching placebo was administered in a 2-sequence crossover design (nested crossover).

DETAILED DESCRIPTION:
Subjects were in-house from Day -2 to Day 20 and were randomized to one of the 2 parallel treatment groups (as part of the blind, both groups received the same number of tablets and capsules at the same timepoints, though some were verum and some were placebo depending on the randomized regimen). Group 1 received a therapeutic and a supra-therapeutic dose of pritelivir plus moxifloxacin placebo. Group 2 received pritelivir placebo as well as one dose of moxifloxacin and one dose of matching placebo in a 2-sequence crossover design (nested crossover). 12-lead electrocardiogram (ECG) triplicates were recorded from the bedside 12-lead ECG on the Days -1, 1, 2, 6, 16, and 17 and were analyzed afterwards in each group for these 6 days of documentation by a blinded reader.

It is of note that Holter ECG data was collected in parallel at Screening to exclude anyone with pre-existing cardiac abnormalities as well as on Days -1, 1, 2, 6, 16, and 17 as a back-up for the bedside 12-lead ECGs.

In Group 1, 32 male and female subjects (at least 12 subjects per sex) received a loading dose of 400 mg pritelivir on Day 1. Afterwards they received 100 mg pritelivir qd from Day 2 to 6 and 400 mg pritelivir qd from Day 7 to 16. Furthermore, these subjects received matching moxifloxacin placebo on the Days 2 and 17.

In Group 2, 32 male and female subjects (at least 12 subjects per sex) receive the respective amounts of tablets of matching pritelivir placebo from Day 1 to Day 16 in Group 2 as verum tablets in Group 1. Furthermore, subjects in Group 2a (16 male and female subjects) received 400 mg moxifloxacin on Day 2 and matching moxifloxacin placebo on Day 17 and subjects in Group 2b (16 male and female subjects) received 400 mg moxifloxacin on Day 17 and matching moxifloxacin placebo on Day 2.

To maintain double-blinding the following measures were needed, and data evaluations generated for Group 1 and Group 2:

* 12-lead ten second ECG triplicates were digitally recorded and analyzed (from the bedside 12-lead-ECG devices) in subjects of both groups on the Days -1, 1, 2, 6, 16 and 17.
* PK samples were collected from subjects of both groups on the Days 1, 6, and 16 for pritelivir and the metabolites AIC090015 and AIC090105 as well as for moxifloxacin on the Days 2 and 17.
* Over-encapsulated moxifloxacin- and matching placebo were used.

ELIGIBILITY:
Inclusion Criteria:

1. Subject had been informed both verbally and in writing about the objectives of the clinical trial, the methods, the anticipated benefits and potential risks and the discomfort to which they may be exposed and had given written consent to participation in the trial prior to trial start and any trial-related procedure.
2. Healthy male and female subjects of any ethnic origin, aged between 18 and 45 years (inclusive). Assessed as healthy based on a Screening examination including medical history, physical examination, blood pressure, pulse rate, ECG assessment, and clinical laboratory results.
3. Male subjects were not planning to father or to donate sperms for in vitro fertilization during the trial and for at least 3 months after dosing of trial medication. Adequate contraception (see below) had to be used during sexual intercourse with women of childbearing potential to make sure the fathering of a child was ruled out during the trial and during the 3 months after dosing of trial medication.

   Women of childbearing potential had to perform adequate contraception. They should also not have donated ova during the trial and for at least 3 months after dosing of trial medication.

   Adequate contraception was defined as a combination of a highly effective method of birth control and additional barrier contraception. Highly effective method of birth control was defined as follows: combined (estrogen and progesterone) oral contraceptives, combined hormonal vaginal rings, hormone implants, hormone injectables, or intrauterine device that needed to be in place for a period of at least 2 months prior to Screening and continue for at least 3 months after dosing of trial medication. Additional barrier contraception (the following methods were allowed: condom of the male, diaphragm with spermicide, cervical cap with spermicide) had to be used for the duration of the trial, defined as from the time of Screening to the End of Trial examination, and for at least 3 months after dosing of trial medication. A single barrier method alone or abstinence alone was not acceptable. Homosexual female subjects who refrained from heterosexual intercourse for at least 3 months prior to Screening could be included without a contraceptive method if they agree to further refrain from heterosexual intercourse until the End of Trial examination, and for at least 3 months after dosing of trial medication.

   Women of non-childbearing potential could be included if surgically sterile (documented complete hysterectomy, supracervical hysterectomy or bi-tubal ligations; partial hysterectomy was not sufficient) or if postmenopausal (who have a history of no menses of at least 24 months at screening and postmenopausal status was confirmed by follicle stimulating hormone [FSH] test at screening).
4. In women, negative serum β-HCG (beta-human chorionic gonadotropin) test at Screening and negative urine β-HCG test on Day -2.
5. Subject agreed to pharmacogenomic blood sampling.
6. Subject had to be willing and able to swallow up to 4 tablets (pritelivir or matching placebo) and 1 capsule (over-encapsulated moxifloxacin or matching placebo) at least twice during the trial.
7. Normal body weight as evidenced by a Body Mass Index (BMI) ≥18.0 and ≤25.0 kg/m2, and a body weight ≥50.0 kg at Screening.
8. Subjects must have a negative test result for HIV-I- and -II-antibody, HBsAg, anti-hepatitis B core antigen (HBc) (IgG + IgM) and anti-hepatitis C virus (HCV) at Screening.
9. Subjects had to have negative urine tests for drugs of abuse (benzodiazepines, opiates, amphetamines, methadone, cocaine, cannabinoids, barbiturates, cotinine) and negative breath alcohol tests at Screening and Admission for the in-house phase (Day -2).
10. Normal triplicate 12-lead ECG measured after 10 minutes in the supine position at screening and on admission on Day -2 showing regular sinus rhythm with a well-defined end of T.
11. Normal 24-hour 12-lead ECG at screening.

Exclusion Criteria:

1. History or current evidence of clinically relevant allergies or idiosyncrasy to drugs or food.
2. History of any moderate or severe allergy or any known allergy to any active or inactive ingredient(s) of moxifloxacin investigational medicinal product (IMP), pritelivir IMP, or their respective matching placebos.
3. Any special dietary requirements that would have prevented the consumption of standardized meals.
4. History or current evidence of any clinically relevant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, hematologic, endocrine, metabolic, neurological, psychiatric, or other disease suspected to influence pharmacokinetics or safety of the IMP.
5. History or any current evidence of a dermatological condition requiring treatment by a general practitioner (GP) or specialist (with the exception of burns, fungal infections, and/or warts).
6. Any other significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the trial, or may bias the result of the trial or the subject's ability to participate in the trial.
7. History of malignancy.
8. Has vital signs consistently outside of normal range at screening or Day -1. Acceptable normal range was as follows:

   * supine heart rate (HR) 40 - 100 bpm (after at least five minutes of supine rest)
   * supine blood pressure (after at least five minutes of supine rest):

     * systolic blood pressure: 90 - 130 mmHg
     * diastolic blood pressure: 40 - 90 mmHg
9. The history or presence of any of the following cardiac conditions: known structural cardiac abnormalities; family history of long QT syndrome; cardiac syncope or recurrent, idiopathic syncope; exercise-related clinically significant cardiac events; known cardiovascular disease.
10. Consistent abnormal interval readings for PR, QRS and QTc intervals (PR <120ms or >210ms, QRS >120ms or QTcF >450ms for males and >470ms for females).
11. Transient fascicular blocks, undue ectopic burden, junctional rhythm and any other ECG findings which may in the opinion of the Investigator make a subject unsuitable for inclusion in this clinical trial.
12. Chronic or clinically relevant acute infections or febrile illness within 5 days prior to administration of the IMP.
13. Clinically relevant abnormalities in serum chemistry, haematology and coagulation parameters, urinalysis. Specifically:

    * Participants with transaminases (AST/ALT) above ULN or total bilirubin x1.5 ULN, at Screening.
    * Hemoglobin below lower limit of normal (LLN) at Screening.
    * Platelet count below LLN at Screening.
    * White Blood Count above upper limit of normal (ULN) at Screening.
    * Participants with urinalysis indicative of underlying infection/pathology at Screening.
14. Magnesium or potassium outside normal range in safety laboratory
15. Subject was lactating or breastfeeding.
16. Subject had received or is planning to receive a COVID-19 vaccination within 4 weeks before first dose administration, or within one week after trial completion. Subject also had to comply with the latest COVID-19 safety measures/testing applicable at the site at that time, for entry into the unit and during in-house stays.

    Note: COVID-19 tests were carried out at regular intervals, prior to entry in the unit and throughout the residential period as per the latest Richmond Pharmacology COVID-19 Infection Control Guidelines and pre-entry algorithms.
17. Use of any medication (incl. over-the-counter medication) within 2 weeks before dosing on Day 1 or within less than 10 times the elimination half-life of the respective drug, or anticipated concomitant medication during the treatment period. Exceptions may be the use of hormonal contraception and hormone replacement therapy as well as single intake of a drug if judged by the Investigators to have no clinical relevance and no relevance for the trial objectives. Eg, limited amounts of paracetamol were allowed to treat painful intercurrent adverse events (eg, headache, migraine).
18. Consumption of methylxanthine-containing beverages or food (coffee, tea, cola, chocolate, "powerdrinks") from 24 h before dosing on Day -1 until discharge.
19. Consumption of alcohol and tobacco products within 48 h prior to admission to the clinic until discharge.
20. Diseases or surgery of the gastrointestinal tract which could have interfered with drug absorption (note: this is not applicable for minor abdominal surgery such as eg, appendectomy and herniotomy).
21. Treatment with an investigational drug within 90 days or 5 half-lives preceding the first dose of trial medication (or as determined by the local requirement, whichever is the longer).
22. Donation of blood or blood products (excluding plasma) within 90 days prior to trial medication administration.
23. Smoking of more than 10 cigarettes/cigars/pipes per day and/or inability to refrain from smoking during confinement.
24. History or clinical evidence of substance and/or alcohol abuse within the 2 years before screening. Alcohol abuse was defined as regular weekly intake of more than 14 units (for both males and females), using the following National Health Service (NHS) alcohol tracker https://www.nhs.uk/oneyou/for-your-body/drink-less/know-your-alcohol-units/
25. Has any finding that, in the view of the Investigator, would compromise the subject's safety requirements or their ability to comply with all the trial requirements.
26. Not able to communicate meaningfully with the Investigator and site staff.
27. Lack of ability or willingness to give informed consent.
28. Participation in an earlier clinical trial with pritelivir.
29. Vulnerable subjects (eg, persons kept in detention).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2022-12-04 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-05-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Richmond Pharmacology Ltd, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Subjects (32 male and female subjects) receive 400 mg pritelivir on Day 1, 100 mg pritelivir from Day 2 to 6 and 400 mg pritelivir from Day 7 to 16.
  Furthermore, these subjects receive moxifloxacin matching placebo on the Days 2 and 17.
  Pritelivir and moxifloxacin placebo: oral administration
- Group 2a: Subjects (16 male and female subjects) received the respective amounts of tablets of matching pritelivir matching placebo on Day 1 to Day 16 in Group 2a as verum tablets in Group1.
  Furthermore, these subjects receive 400 mg moxifloxacin on Day 2 and moxifloxacin matching placebo on Day 17.
  Pritelivir placebo, moxifloxacin and moxifloxacin placebo: oral administration
- Group 2b: Subjects (16 male and female subjects) received the respective amounts of tablets of matching pritelivir matching placebo on Day 1 to Day 16 in Group 2b as verum tablets in Group1.
  Furthermore, these subjects receive moxifloxacin matching placebo on Day 2 and 400 mg moxifloxacin on Day 17.
  Pritelivir placebo, moxifloxacin placebo and moxifloxacin: oral administration
Period: Overall Study
Arm/Group | Group 1 | Group 2a | Group 2b
Started | 32 | 16 | 16
Completed | 32 | 16 | 16
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2a | Group 2b | Total
Number analyzed (Participants) | 32 | 16 | 16 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.5 (4.74) | 27.3 (4.78) | 30.8 (6.23) | 28.2 (5.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 7 | 27
  Male | 20 | 8 | 9 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 2 | 5
  Not Hispanic or Latino | 29 | 16 | 14 | 59
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4 | 0 | 1 | 5
  Black or African American | 2 | 2 | 2 | 6
  White | 20 | 12 | 11 | 43
  Other | 6 | 2 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Effects of Pritelivir on the QTcF Interval (QTc Using Fridericia Correction Method) in Comparison With Placebo in Male and Female Subjects.
Description: Mean QTcF values using the Frederica correction method derived from 12-lead ECGs were used to define the effects of pritelivir in comparison with placebo in male and female subjects.
Time Frame: Day -2 to Day 20
Population: Time course of the drug effect on QTcF: Model based estimates (ECG Set).
Measure: Mean (Standard Deviation); unit: ms
Groups:
- Group 1: Subjects (32 male and female subjects) received 400 mg pritelivir on Day 1, 100 mg pritelivir from Day 2 to 6 and 400 mg pritelivir from Day 7 to 16.
  Furthermore, these subjects received moxifloxacin matching placebo on the Days 2 and 17.
  Pritelivir and moxifloxacin placebo: oral administration
- Group 2a: Subjects (16 male and female subjects) received the respective amounts of tablets of matching pritelivir placebo from Day 1 to Day 16 in Group 2a as verum tablets in Group 1.
  Furthermore, these subjects received 400 mg moxifloxacin on Day 2 and moxifloxacin matching placebo on Day 17.
  Pritelivir placebo, moxifloxacin and moxifloxacin placebo: oral administration
- Group 2b: Subjects (16 male and female subjects) received the respective amounts of tablets of matching pritelivir placebo from Day 1 to Day 16 in Group 2b as verum tablets in Group 1.
  Furthermore, these subjects received 400 mg moxifloxacin on Day 2 and moxifloxacin matching placebo on Day 17.
  Pritelivir placebo, moxifloxacin and moxifloxacin placebo: oral administration.
Arm/Group | Group 1 | Group 2a | Group 2b
Number analyzed (Participants) | 32 | 16 | 16
ms
  Day 1, -1 hour | 402.66 (15.198) | 405.23 (17.208) | 401.94 (16.989)
  Day 1, -40 minutes | 404.55 (15.043) | 408.19 (17.040) | 404.21 (17.782)
  Day 1, -20 minutes | 405.66 (15.781) | 409.10 (15.934) | 405.19 (19.805)
  Day 1, 15 minutes | 405.86 (15.653) | 407.06 (14.679) | 406.23 (16.081)
  Day 1, 30 minutes | 400.94 (14.466) | 403.96 (15.311) | 398.56 (17.347)
  Day 1, 45 minutes | 401.82 (13.891) | 405.48 (17.832) | 402.13 (17.295)
  Day 1, 1 hr | 403.99 (15.280) | 405.69 (17.724) | 403.27 (20.122)
  Day 1, 2 hr | 403.34 (13.638) | 406.42 (16.724) | 404.06 (19.436)
  Day 1, 3 hr | 404.70 (15.006) | 409.08 (17.105) | 403.60 (18.037)
  Day 1, 4 hr | 405.84 (14.719) | 407.63 (16.228) | 403.75 (19,248)
  Day 1, 5 hr | 398.16 (13.577) | 401.54 (16.387) | 401.29 (15.948)
  Day 1, 6 hr | 396.48 (13.705) | 397.56 (15.982) | 396.98 (16.573)
  Day 1, 7 hr | 397.40 (13.037) | 398.69 (17,711) | 396.65 (16.517)
  Day 1, 8 hr | 398.92 (14.727) | 401.81 (16.308) | 397.98 (17.455)
  Day 1, 12 hr | 402.41 (11.990) | 402.63 (15.583) | 402.96 (17.687)
  Day 6, -1 hr | 406.43 (14.456) | 404.94 (13.207) | 404.63 (20.971)
  Day 6, -40 minutes | 405.40 (16.410) | 407.56 (16.518) | 406.60 (18.966)
  Day 6, -20 minutes | 407.01 (16.483) | 405.33 (14.640) | 407.94 (16.662)
  Day 6, 1 hr | 404.76 (15.722) | 406.04 (18.259) | 404.23 (20.257)
  Day 6, 2 hr | 405.93 (15.895) | 404.54 (17.555) | 404.29 (19,128)
  Day 6, 3 hr | 405.34 (17.242) | 404.81 (18.170) | 405.15 (18.768)
  Day 6, 4 hr | 404.73 (16.959) | 406.44 (18.839) | 405.63 (22.097)
  Day 6, 5 hr | 398.04 (13.348) | 396.40 (14.502) | 401.42 (14.800)
  Day 6, 6 hr | 395.97 (14.423) | 396.48 (15.856) | 397.83 (18.350)
  Day 6, 7 hr | 396.82 (14.461) | 396.10 (15.270) | 394.21 (18.831)
  Day 6, 8 hr | 400.02 (13.161) | 397.63 (17.160) | 398.40 (16.213)
  Day 6, 12 hr | 399.09 (12.784) | 396.92 (16.245) | 399.17 (17.726)
  Day 16, -1 hr | 403.56 (15.159) | 405.54 (13.995) | 404.79 (15.734)
  Day 16, -40 minutes | 404.81 (15.116) | 405.54 (17.129) | 405.52 (15.714)
  Day 16, -20 minutes | 405.36 (13.483) | 408.75 (15.479) | 406.38 (14.649)
  Day 16, 1 hr | 403.93 (14.543) | 404.71 (15.240) | 404.88 (15.248)
  Day 16, 2 hr | 404.14 (14.856) | 407.85 (15.755) | 405.15 (18.643)
  Day 16, 3 hr | 405.32 (15.513) | 405.52 (17.318) | 406.83 (16.953)
  Day 16, 4 hr | 405.74 (15.966) | 406.85 (17.257) | 405.38 (16.946)
  Day 16, 5 hr | 398.14 (13.121) | 399.71 (17.031) | 399.56 (14.704)
  Day 16, 6 hr | 395.29 (12.566) | 397.60 (16.424) | 396.04 (16.262)
  Day 16, 7 hr | 396.54 (13.894) | 395.44 (15.874) | 396.42 (17.022)
  Day 16, 8 hr | 400.52 (16.196) | 399.52 (16.536) | 398.46 (15.975)
  Day 16, 12 hr | 398.61 (13.372) | 399.00 (14.569) | 400.23 (15.474)
Statistical Analysis 1: Comparison: Group 1 vs Group 2a vs Group 2b; Test type: Non-Inferiority — Null hypothesis: difference to placebo of change from baseline QTcF ≥ 10 ms; p < 0.05, Mixed Models Analysis; Prediction @ mean max concentration = 0.8, 90% CI 2-sided [-1.3 to 2.9]

ADVERSE EVENTS:
Time Frame: 39 days
Description: Phase 1 trial primarily compares 2 parallel groups: Group 1 receiving pritelivir verum and Group 2 receiving matching pritelivir placebo and moxifloxacin.
  In Group 1 the different pritelivir doses were defined as one intervention with no differentiation between doses, to compare versus pritelivir placebo in Group 2 only. Group 2 (pritelivir placebo arm) was subdivided into subgroups 2a and 2b as subjects received 400 mg moxifloxacin on different days, Day 2 and Day 17, respectively.
Arm/Group | Group 1 | Group 2a | Group 2b
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 20/32 | 10/16 | 10/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=32) | Group 2a (N=16) | Group 2b (N=16)
dizziness (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1)
dizziness postural (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (3) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 5 (5) | 0 (0) | 1 (1)
Neck Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 4 (4) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 5 (6) | 4 (4) | 3 (5)
Erythema ab igne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-11-25): https://cdn.clinicaltrials.gov/large-docs/29/NCT05671029/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-16): https://cdn.clinicaltrials.gov/large-docs/29/NCT05671029/SAP_001.pdf